CLINICAL TRIAL: NCT02689752
Title: A Phase One Open-Label Single-Radiolabeled Dose Study to Investigate the Absorption, Metabolism, And Excretion Of [14C] Fruquintinib (HMPL-013) in Healthy Male Volunteers
Brief Title: A Mass Balance Study to Investigate the Absorption, Metabolism, and Excretion Of [14C] Fruquintinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-013-00CH2
Record Dates: First submitted 2016-02-03; First posted 2016-02-24 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: mass balance; 14C
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fruquintinib (Experimental): fruquintinib suspension, 5 mg （100 mCi）oral taken once
  Interventions: Drug: fruquintinib

INTERVENTIONS:
Drug: fruquintinib — fruquintinib suspension, 5mg ( 100mCi), oral, taken once, fast
  Other Names: HMPL-013

SUMMARY:
This will be an open-label, single-center study to evaluate pharmacokinetics and safety of HMPL-013 in approximately 6 healthy male subjects receiving a single oral 5mg dose of HMPL-013 containing approximately 100 microcuries of [14C] HMPL-013. This study will investigate the absorption, drug biotransformation and mass balance of HMPL-013, seek to identify the compound's major metabolites and supply information for clinical application.

DETAILED DESCRIPTION:
This study will be an open-label, mass balance study of fruquintinib administered orally at 5mg (100mCi). Subjects will be screened for eligibility up to 14 days prior to entry into the study. For study period, subjects will be admitted to the clinical research unit (CRU) on the day before dosing and fast overnight (approximately 10 hours). On the morning of dosing for study period, subjects will receive a single oral dose of 5 mg fruquintinib in the fasted state. Subjects will remain at the CRU for at least 336 hours after administration of study drug for collection of serial blood samples for pharmacokinetic (PK) analysis and safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. A Healthy Male Volunteer between 18 and 40 years of age inclusive;
2. A Body Mass Index (BMI) within the range of 19 to 25 kg/m2 and a total body weight >50kg;
3. Medically normal subjects with no significant abnormal findings at the screening vital signs, physical examination, electrocardiogram (ECG), and laboratory parameters as evaluated by the investigator;
4. Fertile male subjects and their partners are willing to undergo contraception as follows: condom, contraceptive sponge, contraceptive gel, contraceptive diaphragm, intrauterine devices, hormonal contraceptives (oral or injectable), subepidermal contraceptive implant and other contraception methods during the study and until 1 year after taking the dose of investigational product,
5. Subject must voluntarily consent to participate in this study, provide their written informed consent prior to start of any study- specific procedures and be willing to comply with all study procedures.

Exclusion Criteria:

1. Subjects who have a family history of coronary heart disease;
2. Subjects who have a known history of bleeding such as gingival hemorrhage, epistaxis and hemorrhoid bleeding etc.;
3. Subjects have hypertension (Systolic Pressure ≥140 mmHg or Diastolic Pressure ≥90 mmHg);
4. Subjects who are taking, or have taken any drugs that affect metabolism or prescription medication during the screening or within 30 days prior to the screening; Subjects who are taking, or have taken any OTC, herbal remedies or Vitamin during the screening or within 14 days prior to the screening; Subjects who are taking, or have taken any plant extracts like Hypericum Perforatum L. which are not therapeutic but have health function and can affect the absorption and metabolism during the screening or within 3 days prior to the screening; Subjects who have participated in another clinical trial within 2 months prior to the screening;
5. Subjects who are taking, or have taken any drugs which have toxicity to major organs during the screening or within 3 months prior to the screening;
6. Subjects who test positive for nicotine screening or can't quit smoking completely in the study;
7. Subjects who have history or presence of any clinically significant diseases within 3 months prior to the screening;
8. Subjects who have history or presence of gastrointestinal, hepatic, renal diseases or any other known condition that can affect the absorption, distribution, metabolism or excretion of the investigational product;
9. Subjects who have chronic constipation, diarrhea, irritable bowel syndrome or inflammatory bowel disease;
10. Subjects who have hemorrhoids or perianal complications with regular hematochezia;
11. Subjects who have a known history of severe allergic reaction such as drug allergy or had an acute allergic rhinitis or food allergy within 14 days prior to the study medication;
12. Subjects who have donated blood or plasma more than 500ml within 2 months prior to the study medication or more than 50ml within 14 days prior to the study medication;
13. Subjects who have had a positive test for hepatitis B (HBsAg) or hepatitis C (excluded immunization);
14. Subjects who have had a positive test for human immunodeficiency virus (HIV);
15. Subjects who have taken vaccination during the screening or within 6 months prior to the screening;
16. Subjects who have any prior history of substance abuse or treatment (including alcohol) ;
17. Subjects who can't understand the purpose, extent and possible outcomes of the study because of mental disease;
18. Adult subjects who are imprisoned or whose freedom are restricted because of administrative problem or legal issues;
19. Subjects who can't comply with the protocol such as discontinue the follow-up and finish the study according to the protocol;
20. Subjects who are involved in the study design and proceeding such as investigator, pharmacist, clinical research coordinator or other related personnel;
21. Subjects who have any other unsuitable or adverse condition to be determined by the investigator;
22. Subjects who have participated in a radiolabeled clinical trial prior to study medication;
23. Subjects who have been exposed to significant radiation (e.g., x-ray investigation, CT investigation, more than one time radiation exposure in barium meal examination) or whose occupation requires exposure to radiation in the last 12 months.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Total radioactivity on blood, urine and faeces (radiocarbon) following oral suspension [14C]HMPL-013 dosing | Up to 14 days
  Total radioactivity in blood to determine Cmax, Tmax, Half-life, AUC0-t, AUC0-∞ Total radioactivity in urine and faeces at each time interval and cumulative radioactivity (mass balance)

SECONDARY OUTCOMES:
Blood concentrations of HMPL-013 and its metabolites | Up to 14 days
  Blood concentrations of HMPL-013 and its metabolites to determine Cmax, Tmax, Half-life, AUC0-t, AUC0-∞
Mass balance after a single oral dose of [14C] HMPL-013 as generated from recovery of total radioactivity excreted in urine and faeces. | Up to 14 days
Metabolite profililing and identification of metabolites in blood, urine and faeces | up to 14 days
Safety and tolerability parameters, including adverse events (AEs), vital signs, ECGs, and clinical laboratory assessments. | Up to 14 days
  safety will assessed by physical exam, clinical laboratory evaluations and ECGs.

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Su, PHD, Study Director — Hutchison Medipharma Limited
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No